CLINICAL TRIAL: NCT03274050
Title: To Evaluate the Performance and Efficiency of Robotic Surgery in Children and Adults
Acronym: PECRoP
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Intuitive Surgical (Industry); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI16026J; 2017-A01507-46 (Other: IDRCB)
Record Dates: First submitted 2017-07-24; First posted 2017-09-06 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Surgery
Keywords: robot; surgery; pediatry (0-20 years included); adults

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patient group: Surgery with robot - all patients operated in surgery department with indication of robot in the routine care (all specialities).
- control group: Retroperitoneal coelioscopy - patient operated for pyeloplasty - only for pediatry

SUMMARY:
Robotic minimally invasive surgery has been rapidly adopted for a wide variety of surgical procedures in adult patients across a broad spectrum of surgical specialties. This has occurred despite the high costs and uncertain benefits of surgical robots.

In contrast, Children's Hospitals and pediatric surgical disciplines have been much slower to embrace the surgical robot. Many children's hospitals do not even possess a surgical robot, and many of those that do borrow them from the adult operating room within the same medical facility.

Since the first case of robotic minimally invasive surgery in children in 2000, robotic procedures have been slowly adopted by select pediatric surgical specialists.

Advocates of robotic minimally invasive surgical systems add many useful features that include improved dexterity, motion scaling, tremor filtration, greater optical magnification (up to 10x), stereoscopic vision, operator-controlled camera movement, and the elimination of the fulcrum effect when compared to conventional laparoscopy. The wristed laparoscopic instruments used in robotic surgery provide seven degrees of freedom.

For the surgeon, these features may allow for more precise dissection with increased magnification and visibility. The intuitive controls of the robot are purported as providing the ability to perform laparoscopic procedures in an "open" fashion. In pediatric surgical procedures, these technical abilities may have the potential to surpass the physical capabilities of human performance in the tight operative fields encountered in children.

This study aims to evaluate the clinical safety and efficiency in a dedicated multidisciplinary pediatric program and to evaluate the relative cost of robotic surgery

DETAILED DESCRIPTION:
Laparoscopy has been adopted for advantages that include decreased adhesion formation, improved cosmesis, decreased post-operative pain, and shorter recovery times.

The patient benefits of robotic surgery are thought to be essentially the same as conventional laparoscopy: decreased length of stay, decreased blood loss, decreased pain, quicker return to work, and improved cosmetic result through smaller incisions. In pediatric urology, there is evidence that robot-assisted pyeloplasty may be superior to open and laparoscopic approach with decreased length of stay, decreased narcotic use, and decreased operative times.

The overall reported conversion-to-open-procedure rate is low, comparable to the conversion rate in conventional pediatric minimally invasive surgery.

Robotic surgical technology may have a role in pediatric minimal access surgery. Design features of robotic surgical platforms include motion scaling, greater optical magnification, stereoscopic vision, increased instrument tip dexterity, tremor filtration, instrument indexing, operator controlled camera movement, and elimination of the fulcrum effect. These robotic enhancements offer improvements to conventional minimal access surgery, permitting technical capabilities beyond existing threshold limits of human performance for surgery within the spatially constrained operative workspaces in children. There is evidence that a learning curve is encountered when adopting robotic surgery as demonstrated by decreasing operative times as case volumes increased

At a stand-alone pediatric hospital, a robotic platform is often not available. Only a minority of pediatric hospitals have robotic systems given the limited number of procedures performed nationally. This is probably due to the costs of acquiring and maintaining a surgical robot coupled with the tendency for pediatric hospitals to have less income and fewer eligible patients to defray the fixed costs of the platform. A unique situation exists for pediatric surgeons in hospitals affiliated with adult care as robots may be available that are primarily used for adult subspecialties, most often urology. In this setup, the logistics may be difficult and the pediatric team must be flexible and mobile to accommodate the robot.

Robotic surgery has higher costs than open and laparoscopic procedures. This is due to the high costs of purchasing and maintaining a robot, increased operative time, and costs of disposable surgical supplies.

The specificity of this study is to evaluate the clinical safety and efficiency in a dedicated multidisciplinary pediatric program (gastrointestinal surgery, genitourinary surgery, thoracic surgery, ENT, cardiac surgery and microsurgery) and to evaluate the relative cost of robotic surgery.

ELIGIBILITY:
Inclusion Criteria :

* child or adult
* with an indication for a robotic surgery
* non-opposition of patient or non-opposition of parents for minor patient

Exclusion Criteria :

* anatomic or anesthetic contraindication for the mini-invasive surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients operated in surgery department participating of the study with indication of robot in the routine care (all specialities)
Sampling Method: Non-Probability Sample
Enrollment: 16000 (Estimated)
Dates: Start 2018-02-28 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Per and post-surgery complication | 6 months
  per and post-surgery complication (Clavien-Dindo score)

SECONDARY OUTCOMES:
Post-surgery pain with analgesic prescription | 6 months
Resection quality (R0) of oncologic surgery | 6 months
Functional results according to the surgery indication | 6 months
Quality of life (SF-36) | 6 months
  36-items Short Form health survey
Health survey (EQ-5D-5L) | 6 months
  Each dimension in the EQ-5D-5L has five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5)
The Saint-George's hospital Respiratory Questionnaire (SGRQ) | 6 months
  0 indicates best health and 100 indicates worst health
Patient Global Impression of Improvement (PGI-I) | 6 months
  1-question assessment designed to evaluate the patient's impression of improvement since surgery- PGI-I score: 1 = very much better; 2 = much better; 3 = a little better; 4 = no change; 5 = a little worse; 6 = much worse; 7 = very much worse
Frequency and percentage of intervention with robot in each speciality | 6 months
Duration of activity of the operating block | 6 months
Average duration of anaesthesia | 6 months
Average duration of robotic surgery and docking | 6 months
Duration of intervention by speciality (learning curve) | 6 months
Frequency and percentage of conversion to open-procedure | 6 months
Post surgery pain (Evendol pain scale) | 6 months
Prescription of analgesic | 6 months
Duration of hospitalization | 6 months
Cost of robotic surgery by indication, tools and supplies | 6 months
Duration of post surgery work stoppage (activ patient) | 6 months
Duration before returning to normal activity (other patient) | 6 months
Difference in average costs per patients (in €) divided by the difference in post operative complications using the Clavien Dindo scale | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas BLANC, MD; PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Morgane ROUPRET, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker -Enfants Malades, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Franzini S, Querciagrossa S, Brebion M, Consonni D, Blanc T, Orliaguet G. Effect of retropneumoperitoneum on cerebral and renal oxygen saturation during retroperitoneal robotic-assisted laparoscopic pyeloplasty (R-RALP) in a pediatric population: Preliminary results of a prospective observational study using a dedicated anesthetic protocol and Near-InfraRed Spectroscopy. Anaesth Crit Care Pain Med. 2023 Oct;42(5):101234. doi: 10.1016/j.accpm.2023.101234. Epub 2023 Apr 28. PMID 37121359
- [Derived] Vinit N, Vatta F, Broch A, Hidalgo M, Kohaut J, Querciagrossa S, Couloigner V, Khen-Dunlop N, Botto N, Capito C, Sarnacki S, Blanc T. Adverse Events and Morbidity in a Multidisciplinary Pediatric Robotic Surgery Program. A prospective, Observational Study. Ann Surg. 2023 Nov 1;278(5):e932-e938. doi: 10.1097/SLA.0000000000005808. Epub 2023 Jan 23. PMID 36692109
- [Derived] Harte C, Ren M, Querciagrossa S, Druot E, Vatta F, Sarnacki S, Dahmani S, Orliaguet G, Blanc T. Anaesthesia management during paediatric robotic surgery: preliminary results from a single centre multidisciplinary experience. Anaesth Crit Care Pain Med. 2021 Jun;40(3):100837. doi: 10.1016/j.accpm.2021.100837. Epub 2021 Mar 20. PMID 33757915